CLINICAL TRIAL: NCT06852456
Title: A PhaseⅡ/Ⅲ, Randomized, Double-blind, Placebo-controlled Trial to Evaluate QL1706 Perioperative Treatment in Combination With Neoadjuvant Chemotherapy for Locally Advanced, Resectable Esophageal Squamous Cell Carcinoma
Brief Title: QL1706 in Combination With Neoadjuvant Chemotherapy Versus Neoadjuvant Chemotherapy for Locally Advanced, Resectable Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-305
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Resectable Locally Advanced Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 injection combined with chemotherapy (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706)Injection; Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab (QL1706)Injection — PD-1/CTLA-4
Drug: Paclitaxel — Chemotherapy
Drug: Cisplatin — Chemotherapy

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase II/III clinical trial to evaluate the perioperative treatment with QL1706 in combination with neoadjuvant chemotherapy for locally advanced resectable esophageal squamous cell carcinoma. The primary objective of the Phase II is to evaluate the pathological complete response rate of QL1706 perioperative treatment in combination with neoadjuvant chemotherapy for locally advanced resectable esophageal squamous cell carcinoma; the primary objective of the Phase III is to compare event-free survival of QL1706 perioperative treatment in combination with neoadjuvant chemotherapy versus placebo in combination with neoadjuvant chemotherapy for locally advanced resectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1.
* Patients with thoracic esophageal squamous cell carcinoma diagnosed by pathologic histology or cytology and cT1-2N1-3M0 or cT3-4aN0-3M0 according to AJCC/UICC 8th edition.
* Expected to undergo surgery after completion of neoadjuvant therapy and expected to achieve R0 resection.
* Have not receiv any anti-tumor therapy for esophageal cancer.
* Have adequate organ function.

Exclusion Criteria:

* Significant tumor invasion into organs adjacent to the esophageal lesion;
* a history of gastrointestinal bleeding or those with a high bleeding tendency;
* The presence of supraclavicular lymph node metastases;
* the presence of uncontrollable third interstitial fluid;
* poor nutritional status.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate (pCR) as assessed by the investigator; (Phase II stage) | 30 days after operation
  pCR rate was defined as the percentage of subjects with no tumor residue in the primary tumor and regional lymph nodes.
Event-Free Survival (EFS) as assessed by BIRC; (Phase III stage) | up to 5 years
  EFS is defined as the time from randomization (for Phase II: from first dose) to the occurrence of an imaging disease progression/recurrence or death event from any cause, whichever occurs first.